CLINICAL TRIAL: NCT02439372
Title: Assessment of CMV-specific ELISPOT Assay for Predicting CMV Colitis in Patient With Ulcerative Colitis (ACE-UC)
Brief Title: Assessment of CMV-specific ELISPOT Assay for Predicting CMV Colitis in Patient With Ulcerative Colitis
Acronym: ACE-UC
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sung-Han Kim, Associate Professor, Asan Medical Center
Other Study IDs: Report Number 2015-0129
Record Dates: First submitted 2015-04-28; First posted 2015-05-08 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Ulcerative Colitis; Cytomegalovirus Infections; Disease Exacerbation
MeSH Terms: conditions — Colitis, Ulcerative; Cytomegalovirus Infections; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Consequences of latent cytomegalovirus (CMV) infection reactivation on ulcerative colitis flare, as a flare-worsening factor or simple bystander, are debated. Theoretically, CMV-specific cell-mediate immune response will further categorize the patients into high or low risk of CMV colitis. The investigators thus evaluate the usefulness of CMV-specific ELISPOT assay in patient with ulcerative colitis flare to assess the the impact of CMV colitis on ulcerative colitis flare.

DETAILED DESCRIPTION:
Moderate to severe ulcerative colitis patients admitted in Inflammatory Bowel Disease (IBD) center will be enrolled in this study. Eligible patients had active UC with a Mayo score of 6-12 points (moderate or severe disease activity). The investigators will evaluate whether CMV-specific cell-mediated immune response at admission will predict the risk of active cytomegalovirus infection (true pathogen versus bystander).

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe UC require hospitalization
* age 16 or more
* agree with written informed consent

Exclusion Criteria:

* pregnancy
* foreign
* immunosuppressed patients

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Moderate to severe ulcerative colitis (Eligible patients had active UC with a Mayo score of 6-12 points)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
CMV infection | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  CMV colitis (CMV disease involving the colon) was diagnosed by colonic tissue polymerase chain reaction (PCR) or immunohistochemistry (IHC) in accordance with current European guidelines

SECONDARY OUTCOMES:
Viral clearance from colonic mucosa | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Viral clearance from colonic mucosa was diagnosed as negative by immunohistochemistry (IHC) after a ganciclovir treatment
Breakthrough CMV infection | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Breakthrough CMV colitis was diagnosed by newly positive colonic tissue polymerase chain reaction (PCR) or immunohistochemistry (IHC) at the time of second colonic biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Han Kim, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Jung KH, Kim J, Lee HS, Choi J, Jang SJ, Jung J, Kim MJ, Chong YP, Lee SO, Choi SH, Kim YS, Woo JH, Park SH, Yang DH, Ye BD, Yang SK, Kim SH. Clinical Implications of the CMV-Specific T-Cell Response and Local or Systemic CMV Viral Replication in Patients With Moderate to Severe Ulcerative Colitis. Open Forum Infect Dis. 2019 Dec 18;6(12):ofz526. doi: 10.1093/ofid/ofz526. eCollection 2019 Dec. PMID 31893211